CLINICAL TRIAL: NCT00284947
Title: REPLACE: Safety and Efficacy of Basiliximab in Calcineurin Inhibitor Intolerant Long-term Kidney Transplant Recipients Treated With Mycophenolic Acid and Steroids
Brief Title: Safety and Efficacy of Basiliximab in Calcineurin Inhibitor Intolerant Long-term Kidney Transplant Recipients Treated With Mycophenolic Acid and Steroids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CCHI621A2402
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Kidney Transplantation; Adverse Effects
Keywords: Side effects; calcineurin inhibitors; maintenance; basiliximab; Kidney maintenance transplant
MeSH Terms: interventions — Basiliximab; Mycophenolic Acid; Adrenal Cortex Hormones; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Maintenance immunosuppression (Experimental): 40mg Simulect i.v, once every 28 days for 24 weeks (treatment periods)
  * 1g MMF or 720mg EC-MPS p.o twice daily
  * Oral corticosteroids
  Interventions: Drug: basiliximab; Drug: MMF/EC-MPS; Drug: Corticosteroids

INTERVENTIONS:
Drug: basiliximab — 40 mg once every 28 days intravenously for 24 weeks
  Other Names: Simulect
Drug: MMF/EC-MPS — 1g MMF or 720mg EC-MPS p.o twice daily
  Other Names: MPA; Myfortic; Cellcept
Drug: Corticosteroids — Oral corticosteroids, equivalent to prednisone p.o, ≥ 5mg daily or ≥ 10mg on alternate days
  Other Names: Prednisone; Methyl-prednisolone

SUMMARY:
The long-term use of calcineurin inhibitors (CNI) in patients who have received a kidney transplantation is associated with renal dysfunction and hypertension. The study will evaluate the safety and efficacy of replacing the calcineurin inhibitors by using basiliximab at monthly doses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first kidney transplant from a living or deceased donor at least 12 months after transplantation.
* Patients receiving CNI, mycophenolic acid (MPA) and oral corticosteroids.
* Patients who are able to tolerate full dose MPA.
* Patients with glomerular filtration rate (GFR) > 30 mL/min.
* Patients without an acute rejection episode during the preceding 6 months.
* Patients with signs or symptoms of CNI intolerance (renal dysfunction, poor blood pressure control, diabetes, poor lipid control, hyperuricemia and gout, significant hypophosphatemia or hypomagnesemia, gingival hyperplasia, hypertrichosis, etc.) in whom CNI interruption is justified.

Exclusion Criteria:

* Patients with preformed positive skin test against basiliximab
* Patients with preformed panel reactive antibody (PRA) > 10%.
* Signs of active immune process on graft biopsy.
* Patients with multi-organ or second kidney transplant

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
to describe the pharmacokinetics of basiliximab over the 6-month study course and to determine whether serum concentrations remain above CD25 receptor saturation levels | 6 months

SECONDARY OUTCOMES:
to evaluate the risk of sensitization against the chimeric antibody over 6 months | 6 months
to assess the changes in renal parameters after CNI discontinuation | Month 1-6 post trasnplant
to assess the quantifiable changes in vital signs and lab abnormalities possibly related to CNIs | 6 months
to assess semi-quantitatively changes of clinical symptoms possibly related to CNIs | 6 month
to determine the percentage of CD25 positive T cells (CD3) during therapy with Simulect | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, Basel, Switzerland